CLINICAL TRIAL: NCT02488187
Title: Comparison of Preoperative Automated Breast Ultrasound (ABUS) and Magnetic Resonance Imaging (MRI) in Newly Diagnosed Breast Cancer Patients
Brief Title: Comparison of Preoperative ABUS and MRI in Newly Diagnosed Breast Cancer Patients
Acronym: ABUS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Kansas Medical Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: ABUS
Record Dates: First submitted 2015-06-30; First posted 2015-07-02 (Estimated); Last update posted 2017-01-19 (Estimated); Status verified 2016-07

CONDITIONS: Breast Cancer
Keywords: Breast Cancer; MRI; Mammogram; Whole Breast Sonogram; ABUS
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ABUS vs MRI (ultrasound when indicated) (Other): To compare the overall sensitivity and specificity of ABUS versus MRI (and hand-held breast ultrasound when clinically indicated) for the ipsilateral and contralateral breast in newly diagnosed breast cancer patients.
  Interventions: Device: ABUS
- ABUS vs mammography (ultrasound when indicated) (Other): To compare the sensitivity and specificity of ABUS versus mammography (and hand-held breast ultrasound when clinically indicated) for the ipsilateral and contralateral breast in newly diagnosed breast cancer patients when MRI is not performed.
  Interventions: Device: ABUS

INTERVENTIONS:
Device: ABUS — Automated breast ultrasound

SUMMARY:
Comparison of Preoperative Automated Breast Ultrasound (ABUS) and magnetic resonance imaging (MRI) in Newly Diagnosed Breast Cancer Patients.

DETAILED DESCRIPTION:
This is a prospective pilot study investigating the use of Automated Breast Ultrasound in the preoperative evaluation of newly diagnosed breast cancer patients. The Investigator intends to demonstrate that preoperative automated breast ultrasound (ABUS) will provide a relatively inexpensive and well-tolerated alternative to MRI for detection of occult breast cancer missed by mammography and hand-held ultrasound in women with newly diagnosed breast cancer. The research will take place at the University of Kansas Medical Center (KUMC). The research study will be open to newly diagnosed breast cancer patients who present to KUMC with a recommendation for preoperative MRI and who fit all inclusion criteria and have none of the exclusion criteria.

ELIGIBILITY:
Inclusion Criteria:

* Women (age 18-100) undergoing preoperative evaluation at the University of Kansas Cancer Center (KUCC) for a new diagnosis of breast cancer
* Patients with a diagnosis of breast cancer by either core needle biopsy or excisional biopsy.
* Bilateral mammography and hand-held ultrasound (if clinically indicated) performed prior to the MRI and ABUS.
* If a breast MRI is advised and there is no contraindication to MRI, a breast MRI and ABUS will performed at KUCC (Study Arm 1).
* If a breast MRI is not performed, an ABUS exam without MRI will be performed (Study Arm 2).
* The MRI and ABUS exam must be obtained within 2 weeks of each other.

Exclusion Criteria:

* Males
* Pregnant women
* Lactating women
* Patients < 18 and > 100 years of age
* Patients with breast implants

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 115 (Actual)
Dates: Start 2013-04; Primary Completion 2016-07 (Actual); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Measure rate of detection of occult breast cancer by ABUS that was not detected by standard imaging | 1 day
  Rate of detection of occult breast cancer by ABUS, otherwise missed by standard imaging (MRI or mammogram with hand-held breast ultrasound as clinically indicated).

CONTACTS AND LOCATIONS:
Locations (1):
- University of Kansas Cancer Center, Westwood, Kansas, United States